CLINICAL TRIAL: NCT03911453
Title: Window of Opportunity Trial to Evaluate Change in PD-L1 Expression in Triple Negative Breast Tumors in Response to the PARP Inhibitor Rucaparib
Brief Title: Window of Opportunity Trial, PARP Inhibitor Rucaparib Affect on PD-L1 Expression in Triple Negative Breast Tumors
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 30388; 1903397220 (Other: University of Arizona Cancer Center)
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Triple Negative; Breast Tumors; PD-L1; PARP; PARPi; Rucaparib
MeSH Terms: conditions — Breast Neoplasms | interventions — rucaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (rucaparib) (Experimental): Patients will be treated with single agent rucaparib for 3wks and then proceed to surgery. Core-biopsies (at the time of diagnosis) and tumor from the surgical resection will be assessed for change in expression of programmed cell death-1 with ligand (PD-L1) by immunohistochemistry (IHC)
  . Starting Dose 600 mg twice daily Dose Level -1 500 mg twice daily Dose Level -2 400 mg twice daily Dose Level -3 300 mg twice daily
  Interventions: Drug: Rucaparib

INTERVENTIONS:
Drug: Rucaparib — Patients will be treated with single agent rucaparib for 3wks and then proceed to surgery. Core-biopsies (at the time of diagnosis) and tumor from the surgical resection will be assessed for change in expression of PD-L1 by Immunohistochemical assay (IHC).

SUMMARY:
This is a single arm window of opportunity trial conducted in patients with early stage triple negative breast tumors to evaluate if treatment with a Poly(ADP-ribose) polymerase (PARP) inhibitor will increase expression of programmed cell death-1 with ligand (PD-L1) in triple negative breast tumors.

DETAILED DESCRIPTION:
This is a single arm window of opportunity trial conducted in patients with early stage triple negative breast tumors. Patients who are planning to undergo surgery as part of their initial treatment will be eligible for this study. They will be treated with single agent rucaparib for 3 weeks and then proceed to surgery. Core-biopsies obtained at the time of diagnosis and tumor from the surgical resection will be assessed for change in expression of PD-L1 by Immunohistochemical assay (IHC).

ELIGIBILITY:
Inclusion Criteria:

1. Have histologically documented triple negative breast cancer (TNBC) (defined as ER expression ≤10% by IHC, progesterone receptor (PR) expression≤10% by IHC and HER2 0 or 1+ by IHC or Fluorescence in situ hybridization (FISH) ratio <2 or human epidermal growth factor receptor 2 (HER2) gene copy number of <6)
2. Early stage breast cancer (stage I-III) and not be candidate for neoadjuvant chemotherapy
3. Be informed of the investigational nature of the study and all pertinent aspects of the trial
4. Have Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
5. Have the ability to understand and the willingness to sign a written informed consent document in accordance with institutional and federal guidelines
6. Be ≥ 21 years of age
7. Have serum creatinine < 1.5 x institutional upper limit of normal (IULN) or a calculated creatinine clearance ≥ 30ml/min (calculated by Cockcroft Gault equation), bilirubin ≤ 2.0, and an serum glutamic oxaloacetic transaminase (SGOT)/s erum glutamic pyruvic transaminase (SGPT)/alkaline phosphatase ≤ 2.0 x IULN
8. Have adequate bone marrow function (ANC >1000, Platelets >100,000/ml, Hemoglobin >10gm/dL)
9. Women of childbearing potential or male patients of reproductive potential with female partners of childbearing potential must not consider getting pregnant and must avoid pregnancy during the study and for at least 6 months after the last dose of rucaparib. Female and male patients of reproductive potential must practice highly effective methods of contraception with their partners, if of reproductive potential, during treatment and for 6 months following last dose of rucaparib

Exclusion Criteria:

1. Ongoing or prior treatment with a PARPi for breast cancer or other malignancies
2. Receiving concurrent anti-neoplastic therapy for their breast cancer or another malignancy
3. Known documented or suspected hypersensitivity to the components of the study drug or analogs.
4. Pre-existing gastrointestinal disorders or defects (like duodenal stent etc) that would, in the opinion of the investigator, interfere with absorption of rucaparib

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-19 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2021-07-16 (Actual)

PRIMARY OUTCOMES:
Measurement of expression of PD-L1 by IHC via core biopsy. | Six months
  To evaluate change in expression of programmed cell death-1 with ligand (PD-L1) by Immunohistochemistry (IHC) of tissue sample via core biopsy after treatment with single agent PARPi (rucaparib).

SECONDARY OUTCOMES:
Measure change in expression of Ki67 by IHC after treatment with PARPi. | Six months
  Measure change in expression of Ki67 by immunohistochemistry of tissue sample via core biopsy after treatment with single agent Poly(ADP-ribose) polymerase inhibitor (PARPi) (rucaparib).
Measure and quantify change in number of tumor-infiltrating lymphocytes. | Six months
  Measure and quantify change in number of tumor-infiltrating lymphocytes via blood testing.
Measure levels of tumor PARylation in pre- and post-PARPi therapy by IHC. | Six months
  Measure levels of tumor PARylation (the addition of poly-ADP-ribose polymers) in pre- and post-PARPi therapy by immunohistochemistry of tissue sample via core biopsy.
Measure change in expression of programmed cell death-1 with ligand (PD-L1) pre- and post-PARPi therapy in circulating tumor cells (CTCs). | Six months
  Measure change in expression of programmed cell death-1 with ligand (PD-L1) pre- and post-PARPi therapy in circulating tumor cells (CTCs) via blood/plasma collection.
Measure cfDNA mutational expression for homologous recombination deficiency (HRD) and correlate with PD-L1 expression at baseline and change overtime. | Six months
  Measure circulating free DNA (cfDNA) mutational expression for homologous recombination deficiency (HRD) and correlate with PD-L1 expression at baseline and change overtime via blood/plasma collection.

CONTACTS AND LOCATIONS:
Overall Officials: Pavani Chalasani, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Cancer Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No